CLINICAL TRIAL: NCT05065645
Title: A Phase I, Double-blind, Placebo-controlled, Dose-escalation Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Inhaled APN01
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Inhaled APN01 Developed as Treatment for COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apeiron Biologics (Industry)
Collaborators: Apeiron Respiratory Therapies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APN01-01-INHAL
Record Dates: First submitted 2021-08-30; First posted 2021-10-04 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Angiotensin-Converting Enzyme 2; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APN01 (Active Comparator): Angiotensin Converting Enzyme 2: 1.25 mg/ml, 2.5 mg/ml or 5 mg/ml
  Interventions: Drug: Angiotensin Converting Enzyme 2
- NaCl (Placebo Comparator): Sodium Chloride: 0.9% NaCl solution
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Angiotensin Converting Enzyme 2 — SAD: single dose; MAD: dosage 2x daily for 7 days
  Other Names: Inhalation solution
  Arms: APN01
Drug: Sodium chloride — SAD: single dose; MAD: dosage 2x daily for 7 days
  Other Names: Inhalation solution
  Arms: NaCl

SUMMARY:
APN01 is a soluble recombinant form of the human angiotensin-converting enzyme 2 (rhACE2) that is currently under development as a therapy for corona-virus-disease 2019 (COVID-19). By effectively mimicking ACE2 within the body, APN01 is designed to block the SARS-CoV-2 from binding to the ACE2 receptor and infecting cells while at the same time downregulating the renin-aldosterone-angiotensin system (RAAS) to help prevent inflammation and organ injury - critical components involved in the cytokine storm response. ACE2 is the key entry receptor for the SARS-CoV-2. Competitive binding by exogenous angiotensin-converting enzyme 2 (ACE2) may block viral entry, thereby decreasing viral replication in ACE2 expressing organs and protecting the lungs and distal organs from injury induced by SARS-CoV-2.

APN01 has been developed as an IV agent to treat acute lung injury and pulmonary arterial hypertension, and moderate to severe COVID-19 infection. Encouraged by the favorable safety profile of IV APN01, we have developed the nebulized APN01 formulation to deliver the drug directly to the respiratory tract, where the virus is mainly found, decreasing systemic exposure and increasing local pulmonary concentration. APN01 intravenously and as inhalation in preclinical studies has been well tolerated with no overall difference in clinical studies from placebo in human trials to date.

This study will investigate nebulized APN01 safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity before stepping forward in proof-of-concept studies in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females between 18 to 55 years of age, inclusive, at the screening visit.
2. Subject voluntarily agrees to participate in this study and signs an Ethics Committee approved informed consent prior to performing any of the screening visit procedures.
3. Subject is able to understand and is willing to comply with all study requirements, and willing to follow the instructions of the study staff.
4. Women of childbearing potential must have a negative pregnancy test, should not be breastfeeding, and must be willing to use highly effective methods of contraception for at least 1 month before, while participating in this study and until 1 month after the end of the treatment. The following terms of contraception apply:

   4.1. Total abstinence (when this is in line with the preferred and usual lifestyle of the participant). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

   4.2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study intervention. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.

   4.3. Sterilization of male partner (at least 6 months prior to Screening) with post-procedural semen specimen to verify a successful procedure (the report of the male partner will not be collected since the partner is not study participant). For female participants on the study, the vasectomized male partner should be the sole partner for that participant.

   4.4. Placement of an intrauterine device or intrauterine system, or other forms of non-hormonal contraception that have comparable efficacy (failure rate <1%).

   4.5. Women who are postmenopausal are not required to use contraception. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range (FSH > 40 U/ml at Screening) must be used to confirm a postmenopausal state.
5. Male subject must agree to stay abstinent or must use together with his female partner(s) use a form of highly effective contraceptive from the time of signing the informed consent form (ICF) until up to 3 months after receiving the study drug.
6. Nonsmokers (and/or no use of other nicotine products during 1 year before screening visit).
7. Body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive, at the screening visit.
8. Healthy with no clinically significant findings, determined by medical evaluation (medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations) at Screening.
9. Forced expiratory volume in 1 second (FEV1) ≥80%.

Exclusion Criteria:

1. Female subjects who are breastfeeding or female subjects with a positive pregnancy test at the screening visit or admission.
2. Study participant has a history of an anaphylactic reaction to study drug or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
3. Subject has used an investigational drug within 30 days (or 5 half-lives whichever is longer) prior to the first dose of study drug.
4. Subject is on any regular (more than 4 days a week) prescription or nonprescription over the counter medication, topical medications, vitamins, dietary or herbal (occasional use of acetaminophen, paracetamol or ibuprofen allowed).
5. Subject has positive urine test for drugs of abuse at the screening visit or admission.
6. Regular consumption of alcohol within 6 months prior to Screening (> 7 drinks/week for females, > 14 drinks/week for males where 1 drink = 5 ounces [150 ml] of wine or 12 ounces [360 ml] of beer or 1.5 ounces [45 ml] of hard liquor), or use of illicit substances (such as marijuana) within 3 months prior to the screening visit.
7. Subject has positive test for SARS-CoV-2 antigen or real-time RT-PCR, HBsAg, anti-HBc antibodies, HCV antibody, and/or HIV antibody at screening visit.
8. Donation or loss of 450 ml or more of blood within 4 weeks or 250 ml of plasma within 4 weeks prior to initial dosing.
9. Subject has a history or current evidence of a serious and/or unstable cardiovascular, respiratory, gastrointestinal, hematologic, autoimmune, mental or other medical disorder, including cirrhosis or malignancy.
10. Subject has a history of a psychiatric disorder that will affect the subject's ability to participate in the study as determined by the Investigator.
11. Subject has a clinically relevant abnormal ECG.
12. Subject has clinically relevant abnormal laboratory values at the discretion of the Investigator.
13. Subject has hypertension with a mean systolic BP >150 mmHg or mean diastolic BP >100 mm Hg. Screening and admission tests may be repeated once if abnormal.
14. Subject has acute, clinically significant illness within 30 days prior to admission, or any other condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study.
15. Subject is an employee of the clinical research team (any APEIRON Biologics AG or study center employee).
16. Subject is unable to understand the protocol requirements, instructions, study-related restrictions, nature, scope and possible consequences of the clinical study. Subject is unlikely to comply with the protocol requirements, instructions and study-related restrictions, e.g., uncooperative attitude, inability to return for follow-up visits and improbability of completing the clinical study.
17. Subject judged inappropriate as participant for the study by the Investigator for other reasons.
18. Any signs of respiratory tract infection within 6 weeks of screening.
19. Subject previously diagnosed with COVID-19 pneumonia.
20. Presence of acute infection in the preceding 14 days, or presence of fever (> 37.9°C oral or tympanic temperature assessment), or acute symptoms of any severity on the scheduled date of admission.
21. Subject who has a current bacterial, parasitic, fungal, or viral infection; any infection requiring hospitalization or intravenous antibiotics within 6 weeks prior to Screening.
22. Subject has any pathological condition of the oro-laryngeal or respiratory tract that hinders use of nebulizer.
23. Any of the following laboratory abnormalities:

    White blood cells, hemoglobin, platelets, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ±15% outside of normal limits. Alkaline phosphatase (ALP), urea and creatinine above 15% outside of normal limits.
24. Subject has received or plans to receive a coronavirus vaccine, or any other vaccine, within 7 days prior to the first dose of study drug or during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Adverse events | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Incidence of adverse events (AEs), serious AEs (SAEs), study withdrawals due to AEs, adverse drug reactions (ADRs), and all-cause death,
Vital signs: Supine blood pressure assessed by systolic and diastolic blood pressure in mmHg | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Systolic and diastolic blood pressure in mmHg
Vital signs: Resting pulse rate measured in beats per minute | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Resting pulse rate measured in beats per minute
Vital signs: Body temperature assessed contactless via TriTemp thermometer in degree C | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Body temperature measured in degree C
Vital signs: Respiratory rate measured in breaths/min | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Respiratory rate measured in breaths/min
Vital signs: Peripheral oxygen saturation (SaO2) measured in % | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Peripheral oxygen saturation (SaO2) measured in %
Clinical laboratory tests: Clinically significant changes of hematology, clinical chemistry and coagulation assessed via blood sample collection | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Clinically significant changes of hematology, clinical chemistry, coagulation and urinalysis assessed via blood sample collection
Clinical laboratory tests: Clinically significant changes of urinalysis measurement assessed via urin collection | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Clinically significant changes of urinalysis measurement assessed via urin collection
Physical examination: Abnormal findings of the general appearance | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of general appearance
Physical examination: Abnormal findings of the ears | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the ears
Physical examination: Abnormal findings of the nose | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the nose
Physical examination: Abnormal findings of the head | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the head
Physical examination: Abnormal findings of the eyes | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the eyes
Physical examination: Abnormal findings of the dermatologic system | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the dermatologic system
Physical examination: Abnormal findings of the mouth/throat/neck | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the mouth/throat/neck
Physical examination: Abnormal findings of the thyroid | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the thyroid
Physical examination: Abnormal findings of the lymph nodes | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the lymph nodes
Physical examination: Abnormal findings of the respiratory system | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the respiratory system
Physical examination: Abnormal findings of the cardiovascular system | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the cardiovascular system
Physical examination: Abnormal findings of the gastrointestinal system | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the gastrointestinal system
Physical examination: Abnormal findings of the extremities | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the extremities
Physical examination: Abnormal findings of the musculoskeletal system | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the musculoskeletal system
Physical examination: Abnormal findings of the neurologic system | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the neurologic system
Physical examination: Abnormal findings of the psychiatric system | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Abnormal findings of the psychiatric system
Heart function: QT interval corrected for heart rate (QTc) (Bazett's correction [QTcB]) in msec assessed via Twelve lead ECG | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Twelve lead ECG: QT interval corrected for heart rate (QTc) (Bazett's correction [QTcB]) measured in msec
Pulmonary function assessed via Forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) measured in L by spirometry | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) measured in L
Pulmonary function assessed via Peak expiratory flow (PEF) measured in L/s by spirometry | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Peak expiratory flow (PEF) measured in L/s
Pulmonary function assessed via FEV1/FVC ratio measured in % by spirometry | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  FEV1/FVC ratio measured in %
Pulmonary function assessed via Total lung capacity (TLC) and Residual volume (RV) measured in L by body plethysmography | SAD cohort: 2 weeks, MAD cohort: 3 weeks
  Total lung capacity (TLC) and Residual volume (RV) measured in L
Fractional Exhaled Nitric Oxide (FeNO) levels measured in parts per billion (ppb) - in MAD cohort only | MAD cohort: 3 weeks
  Fractional Exhaled Nitric Oxide (FeNO) levels measured in parts per billion (ppb)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Bauer M, Jorda A, Al-Jalali V, Wolfl-Duchek M, Bergmann F, Nussbaumer-Proll A, Steindl A, Gugenberger R, Bischof S, Wimmer D, Idzko M, Zeitlinger M. Phase I dose-escalation study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of an inhaled recombinant human ACE2. ERJ Open Res. 2024 Feb 19;10(1):00567-2023. doi: 10.1183/23120541.00567-2023. eCollection 2024 Jan. PMID 38375429
- [Derived] Shoemaker RH, Panettieri RA Jr, Libutti SK, Hochster HS, Watts NR, Wingfield PT, Starkl P, Pimenov L, Gawish R, Hladik A, Knapp S, Boring D, White JM, Lawrence Q, Boone J, Marshall JD, Matthews RL, Cholewa BD, Richig JW, Chen BT, McCormick DL, Gugensberger R, Holler S, Penninger JM, Wirnsberger G. Development of an aerosol intervention for COVID-19 disease: Tolerability of soluble ACE2 (APN01) administered via nebulizer. PLoS One. 2022 Jul 11;17(7):e0271066. doi: 10.1371/journal.pone.0271066. eCollection 2022. PMID 35816490